CLINICAL TRIAL: NCT01000766
Title: Identification of New Biomarkers of Drug Induced Liver Injury
Brief Title: Identifying Changes in Blood (Potential Biomarkers) in Individuals With Drug-Induced Liver Injury
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 50KR10957
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Drug Induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute drug-induced liver injury

SUMMARY:
The purpose of this study is to try to develop new blood tests that may help doctors identify if a drug is hurting a person's liver.

DETAILED DESCRIPTION:
Our hypothesis is that there are liver-specific particles, called mRNA, that are identifiable in a person's blood sample during liver injury caused by some drugs. The purpose of this study is to try to develop new blood tests that may help doctors identify if a drug is hurting a person's liver, perhaps early in the process before significant injury or illness have occurred.

ELIGIBILITY:
Inclusion Criteria:

* ALT > 200 IU/L at presentation to UNC Hospitals
* Drug induced liver injury considered likely by admitting medical staff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in emergency rooms or inpatients at the University of North Carolina Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Watkins, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States